CLINICAL TRIAL: NCT02259218
Title: Biomarker Discovery for Toxicity and Survival in Radiation Oncology: An Integrative Molecular-Clinical Approach
Brief Title: Metabolomic and Epigenetic Profiling of Bodyfluids From Lung and Brain Cancer Receiving Radiation Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Arnab Chakravarti, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-11108; NCI-2014-01575 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-09-11; First posted 2014-10-08 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Adult Brain Tumor; Lung Cancer; Radiation Toxicity
Keywords: Biomarker; Radiation
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, urine, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative: Prospectively collected blood, urine, and tissue samples are analyzed for potential predictive biomarkers via metabolomic and other molecular profiling.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies metabolomic and other molecular profiling to identify predictive biomarkers for radiation toxicity and survival in patients with lung or brain cancers receiving radiation therapy. Studying samples of blood, urine, and tissue from patients with lung or brain cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer and predict which patients are at higher risk for developing radiation side effects and how well patients will respond to radiation treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Metabolomic and epigenetic urine and blood profiles of patients undergoing radiation therapy for lung cancer associated with the development of radiation pneumonitis.

II. Metabolomic and epigenetic urine and blood profiles of patients undergoing radiation therapy for brain cancer associated with the development of radiation necrosis.

SECONDARY OBJECTIVES:

I. Metabolomic and epigenetic urine, blood, and tissue profiles of patients undergoing radiation therapy for lung and brain cancer associated with survival.

OUTLINE:

Collected blood, urine, and tissue samples are analyzed for biomarkers via metabolomic and epigenetic profiling using mass spectrometry, array, and sequencing-based technology.

ELIGIBILITY:
Inclusion Criteria:

* Consultation with the Radiation Oncology department of the Ohio State University (OSU) Comprehensive Cancer Center
* The following diagnoses will be included: malignant neoplasm of the brain; primary malignant neoplasm of trachea bronchus and lung; primary malignant neoplasm of the cervix uteri and primary malignant neoplasm the prostate

Exclusion Criteria:

* Being an inmate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with lung, brain, prostate or cervical cancer that are being treated with radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Potential predictive biomarkers for the development of radiation pneumonitis for lung cancer patients | Baseline
  For each biomarker, linear mixed model (with group and time interaction and repeated measurement for each patient over time) on the log-transformed expression level will be used to detect if it is differentially expressed after controlling for the effects of the co-variates (such as age, disease status, and treatment details).
Potential predictive biomarkers for the development of radiation necrosis for brain cancer patients | Baseline
  For each biomarker, linear mixed model (with group and time interaction and repeated measurement for each patient over time) on the log-transformed expression level will be used to detect if it is differentially expressed after controlling for the effects of the co-variates (such as age, disease status, and treatment details).

SECONDARY OUTCOMES:
Biomarkers that are prognostically significant on disease free or overall survival, identified using the survival analysis | Baseline
  Kaplan Meier analysis and logrank test to identify biomarkers that are prognostically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Chakravarti, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu